CLINICAL TRIAL: NCT05906563
Title: Clinical and Radiographic Evaluation of Melatonin and Metformin Loaded Nanoparticles in the Treatment of Periodontal Intra-bony Defects: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Melatonin and Metformin Loaded Nanoparticles in the Treatment of Periodontal Intra-bony Defects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Amira ragab (Other)
Responsible Party: Sponsor-Investigator, Amira ragab, BDS, clinical demonstrator, Oral Medicine, Periodontology, Diagnosis and Oral Radiology Department, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A06011122
Record Dates: First submitted 2023-03-14; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Bone Loss in Jaw
Keywords: nanoparticles; melatonin; metformin; intra-bony defect
MeSH Terms: interventions — Metformin; Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: triple blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- melatonin loaded nanoparticle (test group) (Active Comparator): 13 patients will be treated with melatonin loaded nanoparticle gel as adjunct to scaling and root planning .it will be applied once weekly for four weeks.
  Interventions: Drug: Melatonin gel; Procedure: scaling and root planning
- melatonin and metformin loaded nanoparticle (test group) (Active Comparator): 13 patients will be treated with melatonin and metformin loaded nanoparticle gel as adjunct to scaling and root planning .It will be applied once weekly for four weeks.
  Interventions: Drug: Metformin and melatonin gel; Procedure: scaling and root planning
- placebo gel (control group) (Placebo Comparator): 13 patients will be treated with placebo gel as adjunct to scaling and root planning .It will be applied once weekly for four weeks.
  Interventions: Drug: placebo gel; Procedure: scaling and root planning
- no gel (control group) (Other): 13 patients will be treated with only scaling and root planning ..
  Interventions: Procedure: scaling and root planning

INTERVENTIONS:
Drug: Melatonin gel — local application of Melatonin gel into the periodontal pocket using a syringe with a blunt cannula until the pocket will be completely filled. It will be applied once weekly for four weeks. After insertion of the local drug delivery system, the region will be secured with a periodontal pack
  Arms: melatonin loaded nanoparticle (test group)
Drug: Metformin and melatonin gel — local application of Metformin and melatonin gel into the periodontal pocket using a syringe with a blunt cannula until the pocket will be completely filled. It will be applied once weekly for four weeks. After insertion of the local drug delivery system, the region will be secured with a periodontal pack
  Arms: melatonin and metformin loaded nanoparticle (test group)
Drug: placebo gel — Local application of empty nanoparticles gel into the periodontal pocket using a syringe with a blunt cannula until the pocket will be completely filled. It will be applied once weekly for four weeks. After insertion of the local drug delivery system, the region will be secured with a periodontal pack.
  Arms: placebo gel (control group)
Procedure: scaling and root planning — full mouth supra- and subgingival scaling and root planning will be performed, and all periodontitis patients will be treated with ultrasonic tips and Gracey curettes for meticulous removal of subgingival and supragingival plaque and calculus.

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of local delivery of melatonin and metformin loaded nanoparticle gel as adjunct to scaling and root planning (SRP) in the treatment of periodontal intra bony defect.

fifty two healthy patients(n=52) with at least one periodontal intra-bony defect will be included in the study, all selected patients will be motivated about the benefit of plaque control and periodontal treatment . The participant will be selected from outpatient clinic of the Department of Oral Medicine and Periodontology , Faculty of dentistry, Mansoura University . The participant will be classified into four groups :group I and II are test groups but group III and IV are control groups .Patients in group I will be treated with melatonin loaded nanoparticle gel while in group II will be treated with melatonin and metformin loaded nanoparticles which will be applied weekly for four weeks after SRP had been completed and group III will be treated with placebo gel while group IV will be treated with only scaling and root planning.

ELIGIBILITY:
Inclusion Criteria:

* patients with at least one intra-bony defect diagnosed clinically and radiographically

Exclusion Criteria:

* Patients with systemic diseases.
* Pregnant and lactating females.
* Smokers and tobacco chewers.
* History of antibiotic and periodontal therapy in the last 3 months.
* Patients not compliant with oral hygiene procedures.
* Patients with a known or suspected allergy to the melatonin or metformin.
* Individuals on systemic drug affecting metabolic bone diseases and medically compromised patients.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Radiographic assessment | all the parameter will be evaluated after 6 months
  all the radiographic parameters will be measured on cone beam computed radiography (CBCT) .The depth of intra bony defect will be measured from cemento enamel junction(CEJ) to base of the defect (BD).The Height of the defect from CEJ to the crest of bone adjacent to the defect and the width of the defect will be from highest point of alveolar crest to dental root adjacent to defect .

SECONDARY OUTCOMES:
plaque index according to Silness P.Loe H 1964 | 6 months
  Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3. The scores from the four areas of the tooth are added and divided by four in order to give the plaque index for the tooth with the following scores and criteria:
  The Plaque Index System
  0 No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2. Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.

OTHER OUTCOMES:
Gingival bleeding index(GBI - Ainamo & Bay, 1975) | 6 months
  is performed through gentle probing of the orifice of the gingival crevice. If bleeding occurs within 10 seconds a positive finding is recorded and the number of positive sites is recorded and then expressed as a percentage of the number of sites examined.
Probing Pocket depth (PPD) | 6 months
  Is measured from free gingival margin to base of the pocket
Clinical Attachment level (CAL) | 6 months
  Is measured from cementoenamel junction to base of the pocket

CONTACTS AND LOCATIONS:
Overall Officials: Amira R AL-Agooz, Principal Investigator — Mansoura University, Faculty of Dentistry
Locations (1):
- Amira R agab AL-agooz, Al Mansurah, Dakhlia, Egypt